CLINICAL TRIAL: NCT03728400
Title: Follow-up of Malnutrition Screening in Neurovascular Intensive Care Unit
Brief Title: Follow-up of Malnutrition Screening in USINV
Acronym: DENUTRITION
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: DENUTRITION USINV
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients in neurovascular intensive care: During the patient's hospitalization in neurovascular intensive care unit, the doctor will propose to the patient to take part in this study. If the patient agree, this search will not change the patient's usual support and will not involve any further review.

SUMMARY:
This aim of the study is to set up a procedure for screening for undernutrition in the neurovascular intensive care unit. This screening procedure follows a specific work concerning undernutrition in thrombolyzed patients (NCT03303820). This work was motivated by the fact that, despite a high frequency of undernutrition in the hospital (at least 30% of patients), undernutrition in neurovascular unit is studied very little. A cohort of thrombolysed patients in 2014 was studied retrospectively. Patients malnourished at the entrance had a non-significant, less good recovery of their stroke (+ 1 Rankin score point at 3 months in malnourished patients at the entrance).

DETAILED DESCRIPTION:
The main objective of this project is to assess, prospectively, the frequency of undernutrition at the entrance to the neurovascular intensive care unit and to evaluate the implementation of the undernutrition screening procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 70 years
* Patient hospitalized in Neurovascular Intensive care Unit following a stroke (infarction or cerebral hematoma)
* Francophone patient

Exclusion Criteria:

* Patient hospitalized in Neurovascular Intensive care Unit following a transient ischemic attack
* Patient whose age ≤ 70 years
* Patient hospitalized in Neurovascular Intensive care Unit for another reason than neurovascular disease
* Patient opposing the use of his data

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients hospitalized in Neurovascular Intensive care Unit following a stroke
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
frequency of undernutrition at the entrance | Day 1
  The primary endpoint is the number of patients who have had an assessment of their nutritional status, that is, for whom undernutrition is detected according to the terms proposed in the undernutrition screening procedure: search for previous quantified weight loss, input BMI, albuminemia.

SECONDARY OUTCOMES:
Modified Rankin scale | 3 months
  The Rankin score will be performed in post stroke consultation, 3 months after inclusion. Rankin scale: 0 no symptoms, 1 No significant disability. Able to carry out all usual activities, despite some symptoms, 2 Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities, 3 Moderate disability. Requires some help, but able to walk unassisted, 4 Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted, 5 Severe disability. Requires constant nursing care and attention, bedridden, incontinent
Recurrence rate of ischemic or haemorrhagic stroke | 3 months
  The recurrence of stroke will be collected during the post stroke consultation, 3 months after inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Marie P BRUANDET, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided